CLINICAL TRIAL: NCT01844024
Title: Task Sharing to Improve Post Abortion Care at District Health Care Level- Trial in Uganda
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Makerere University (Other)
Responsible Party: Principal Investigator, Kristina Gemzell Danielsson, Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Tasksharing PAC
Record Dates: First submitted 2013-04-15; First posted 2013-05-01 (Estimated); Last update posted 2014-08-29 (Estimated); Status verified 2014-08

CONDITIONS: Pregnancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- misoprostol by midwife (Other): Women with incomplete abortion is diagnosed and treated with misoprostol by midwife
  Interventions: Other: misoprostol by midwife
- Misoprostol by physician (No Intervention): Women with incomplete abortion is diagnosed and treated with misoprostol by physician

INTERVENTIONS:
Other: misoprostol by midwife — Women with incomplete abortion is diagnosed and treated with misoprostol by midwife
  Arms: misoprostol by midwife

SUMMARY:
Uganda is one of the countries with highest fertility rate in the world, 6.7 children per women. It is estimated that 56 percent of all pregnancies are unintended and the contraceptive prevalence rate in Uganda is 23 percent. Unwanted pregnancy is common and induced abortion is illegal. Unsafe abortion is responsible for significant morbidity and mortality among women in Uganda. Almost 40% of admissions to emergency obstetric care units in Uganda due to unsafe abortion is reported and considered high in international comparison. Studies have revealed that trained midlevel providers can deliver safe post abortion care (PAC) for incomplete abortion and use manual vacuum aspiration. The prostaglandin E1 analogue misoprostol has been shown to be an effective tool in the treatment of incomplete abortions. This option is so far under-used in developing countries, especially outside the larger hospitals and private clinics. One significant limiting factor in providing safe PAC is the lack of providers. So far technical training has been mainly limited to physicians. The long-term goal of this project is to provide evidence based information that will contribute to the development of strategies to increase women's access to high level post- abortion care at primary health care level provided by midlevel providers in Uganda. A task shift to midlevel provider in providing treatment of incomplete abortion will increase access to safe PAC and is a key to Millenium Development Goal 5. Misoprostol treatment of incomplete abortion remains underused and in accessible to a majority of women in Uganda because national regulations restricts its prescription and supervision to doctors. However, the safety of misoprostol treatment should make it amenable to provision by midlevel providers. Training of midlevel providers in misoprostol treatment of incomplete abortion will support task shifting in places where doctors are costly and scarce. By evaluating the effectiveness of mid-level providers (midwives); administering misoprostol treatment of incomplete abortion the project is attempting to contribute to the reduction of maternal mortality and morbidity and safeguard high quality of post-abortion care. A direct economic impact can also be expected due to reduced treatment costs of complications from unsafely induced abortion and incomplete abortions. The involvement of midlevel providers in medical treatment of incomplete abortion has previously not been systematically evaluated in African primary health care setting.

ELIGIBILITY:
Inclusion Criteria:

* bleeding and contractions during pregnancy

Exclusion Criteria:

* women with known allergy to misoprostol,
* a uterine size more than 12 weeks of gestation,
* suspected ectopic pregnancy,
* unstable hemodynamic status and chock,
* signs of pelvic infection and/or sepsis.

Min Age: 15 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1010 (Actual)
Dates: Start 2013-04; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Complete abortion | 14 days
  The clinical assessments of the main outcome are: (i) Physical examination (pulse, blood pressure and temperature); (ii) Pelvic examination that includes examination of size of the uterus (external genitalia, speculum examination, bimanual examination).

SECONDARY OUTCOMES:
bleeding | 14 days
  Measurements of secondary outcomes are: (i) symptom diary card used by women to assess daily bleeding . The intensity of bleeding will be self-reported by the women in relation to normal menstrual bleeding (categorised 1=much less than up to 5= much heavier than).
pain | 14 days
  Measurements of secondary outcomes are: (i) symptom diary card used by women to assess pain. Pain reported using visual analogue scale (VAS). before any use of analgesia.
acceptability | 14 days
  Standardized questionnaires will be used to collect information about women's acceptability and experiences of the treatment and time spent on travelling and on clinical visits following treatment.
un-scheduled visits | 14 days
  Standardized questionnaires will be used to collect information about women's time spent on travelling and on clinical visits following treatment.

OTHER OUTCOMES:
contraceptive up take | 14 days
  Standardized questionnaires will be used to collect information about women's pre and post contraceptive uptake.

CONTACTS AND LOCATIONS:
Overall Officials: Josaphat Byamugisha, MD, PhD, Principal Investigator — Makerere University
Locations (1):
- Mulago Hospital, Kampala, Uganda

REFERENCES:
- [Derived] Ghosh J, Papadopoulou A, Devall AJ, Jeffery HC, Beeson LE, Do V, Price MJ, Tobias A, Tuncalp O, Lavelanet A, Gulmezoglu AM, Coomarasamy A, Gallos ID. Methods for managing miscarriage: a network meta-analysis. Cochrane Database Syst Rev. 2021 Jun 1;6(6):CD012602. doi: 10.1002/14651858.CD012602.pub2. PMID 34061352
- [Derived] Cleeve A, Byamugisha J, Gemzell-Danielsson K, Mbona Tumwesigye N, Atuhairwe S, Faxelid E, Klingberg-Allvin M. Women's Acceptability of Misoprostol Treatment for Incomplete Abortion by Midwives and Physicians - Secondary Outcome Analysis from a Randomized Controlled Equivalence Trial at District Level in Uganda. PLoS One. 2016 Feb 12;11(2):e0149172. doi: 10.1371/journal.pone.0149172. eCollection 2016. PMID 26872219
- [Derived] Klingberg-Allvin M, Cleeve A, Atuhairwe S, Tumwesigye NM, Faxelid E, Byamugisha J, Gemzell-Danielsson K. Comparison of treatment of incomplete abortion with misoprostol by physicians and midwives at district level in Uganda: a randomised controlled equivalence trial. Lancet. 2015 Jun 13;385(9985):2392-8. doi: 10.1016/S0140-6736(14)61935-8. Epub 2015 Mar 27. PMID 25817472